CLINICAL TRIAL: NCT05756192
Title: An Educational Video's Impact on Knowledge About HPV Vaccination and Cervical Cancer Screening Among Hispanic Patients: a Randomized Control Trial
Brief Title: Educational Video's Impact on Knowledge Regarding Cervical Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Stephanie Wang, Principal Investigator, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCR224166
Record Dates: First submitted 2023-01-30; First posted 2023-03-06 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Human Papilloma Virus; Cervical Dysplasia
Keywords: cervical cancer screening; pap smear; HPV vaccination
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Care providers will be masked as we do not want bias to impact provider counseling at time of visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video and physician counseling arm (Experimental): This groups will complete a pre survey and will then watch the 10-minute educational video on cervical cancer screening and prevention prior to seeing their provider. Patients will then see the provider and will complete a post survey following appointment.
  Interventions: Other: Educational video
- Physician counseling arm (No Intervention): This group will complete a pre survey and will then see their provider. Following provider visit patients will complete a post survey.

INTERVENTIONS:
Other: Educational video — Intervention is a 10-minute animated video that explains cervical cancer screening and prevention.
  Arms: Video and physician counseling arm

SUMMARY:
The researchers will be conducting a prospective randomized trial where the researchers will be introducing an educational video to see whether there is an increase in knowledge scores surrounding cervical cancer, cervical cancer screening, and prevention with HPV vaccinations.

DETAILED DESCRIPTION:
The researchers are conducting a single-blinded randomized controlled trial. All patients who meet exclusion criteria will be recruited at the time of their visit where a Pap smear will be collected at an ob/gyn clinic. If patients agree to participate in the study, they will be randomized into one of two arms. A control arm or an interventional arm. The control arm just includes physician counseling regarding cervical cancer screening/prevention, while the interventional arm includes patient's watching a video on cervical cancer screening/prevention as well as physician counseling. Patient will be administered a survey before and after to assess knowledge and satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Hispanic patients
* Between age 21-65 y/o
* Receiving pap smear during clinic appointment

Exclusion Criteria:

* Non-female patients
* Non-Hispanic patients
* Age less than 21
* Age greater than 65
* not receiving pap smear

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Pre Knowledge score | Will be measured immediately before the appointment.
  Knowledge scores regarding cervical cancer screening and prevention. This will be scored as percentage correct out of 13 questions.
Post knowledge score | Will be measured immediately after the appointment.
  Knowledge scores regarding cervical cancer screening and prevention. This will be scored as percentage correct out of 13 questions.

SECONDARY OUTCOMES:
Post Satisfaction scores | Will be measured immediatley after the provider visit and/or administration or video based educational tool (if randomized to the intervention line).
  Satisfaction scores regarding intervention and appointment. Satisfaction questions will be scored on Likert scale from 1-5 with 5 being most satisfied and 1being the least sat

CONTACTS AND LOCATIONS:
Locations (1):
- Stephanie Wang, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olusola P, Banerjee HN, Philley JV, Dasgupta S. Human Papilloma Virus-Associated Cervical Cancer and Health Disparities. Cells. 2019 Jun 21;8(6):622. doi: 10.3390/cells8060622. PMID 31234354
- [Background] Gibb RK, Martens MG. The impact of liquid-based cytology in decreasing the incidence of cervical cancer. Rev Obstet Gynecol. 2011;4(Suppl 1):S2-S11. PMID 21617785
- [Background] Joura EA, Giuliano AR, Iversen OE, Bouchard C, Mao C, Mehlsen J, Moreira ED Jr, Ngan Y, Petersen LK, Lazcano-Ponce E, Pitisuttithum P, Restrepo JA, Stuart G, Woelber L, Yang YC, Cuzick J, Garland SM, Huh W, Kjaer SK, Bautista OM, Chan IS, Chen J, Gesser R, Moeller E, Ritter M, Vuocolo S, Luxembourg A; Broad Spectrum HPV Vaccine Study. A 9-valent HPV vaccine against infection and intraepithelial neoplasia in women. N Engl J Med. 2015 Feb 19;372(8):711-23. doi: 10.1056/NEJMoa1405044. PMID 25693011
- [Background] Henk HJ, Insinga RP, Singhal PK, Darkow T. Incidence and costs of cervical intraepithelial neoplasia in a US commercially insured population. J Low Genit Tract Dis. 2010 Jan;14(1):29-36. doi: 10.1097/LGT.0b013e3181ac05e9. PMID 20040833
- [Background] Lichter K, Krause D, Xu J, Tsai SHL, Hage C, Weston E, Eke A, Levinson K. Adjuvant Human Papillomavirus Vaccine to Reduce Recurrent Cervical Dysplasia in Unvaccinated Women: A Systematic Review and Meta-analysis. Obstet Gynecol. 2020 May;135(5):1070-1083. doi: 10.1097/AOG.0000000000003833. PMID 32282601
- [Background] Akinlotan M, Bolin JN, Helduser J, Ojinnaka C, Lichorad A, McClellan D. Cervical Cancer Screening Barriers and Risk Factor Knowledge Among Uninsured Women. J Community Health. 2017 Aug;42(4):770-778. doi: 10.1007/s10900-017-0316-9. PMID 28155005
- [Background] Rahman S, Kripalani S, Keegan E, Sparks A, Amdur R, Moawad G, Sheth S, Klebanoff J. An educational video's impact on the induction of labor experience: a randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Jan;4(1):100495. doi: 10.1016/j.ajogmf.2021.100495. Epub 2021 Sep 24. PMID 34571210
- [Background] Pallett AC, Nguyen BT, Klein NM, Phippen N, Miller CR, Barnett JC. A randomized controlled trial to determine whether a video presentation improves informed consent for hysterectomy. Am J Obstet Gynecol. 2018 Sep;219(3):277.e1-277.e7. doi: 10.1016/j.ajog.2018.06.016. Epub 2018 Jun 28. PMID 29959929
- [Derived] Wang SM, Rahman S, Salinas M, Castro J, Aldous A, Huerta E, Chappell NP. Impact of educational video on cervical cancer knowledge in hispanic patients: A randomized trial. Patient Educ Couns. 2025 Sep;138:109202. doi: 10.1016/j.pec.2025.109202. Epub 2025 Jun 6. PMID 40483901